CLINICAL TRIAL: NCT04368065
Title: Registry to Study Factors That May Impact COVID-19 Occurrence and Severity
Brief Title: COVID-19 Active Research Experience (CARE)
Status: Completed | Type: Observational
Sponsor: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IQVIA_COVIDREGISTRY_2020
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 Active Research Experience (CARE) is an observational, direct-to-participant, web-based, longitudinal study of adults with COVID-19 or COVID-19 like illness or who were vaccinated against COVID-19 to better understand risk factors, symptoms, and treatments for COVID-19 illness and vaccine safety and effectiveness.

DETAILED DESCRIPTION:
This is an observational, direct-to-participant, web-based, longitudinal study of adults with COVID-19 or COVID-19 like illness to better understand risk factors, symptoms, and treatments for COVID-19 illness and vaccine safety and effectiveness. Upon consent and enrollment, participants will complete an initial baseline survey reporting their demographics, relevant medical history, testing, vaccination, symptoms, use of prescription medications as well as use of supplements and other factors. The study follow-up period is 12 months. During the first month of follow-up participants will be invited to complete a symptom diary weekly to gauge symptom progression and severity and to provide updates on pharmaceutical and non-pharmaceutical interventions as well as healthcare encounters. Reporting will then reduce to monthly for Month 2 through 12.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Currently living in the US or UK
* Have regular access to a computer, smartphone or tablet and sufficient internet to support registry demands (note: this registry is designed to operate well even in regions with low bandwidth)
* Willing and able to provide informed consent
* Willing and able to follow the procedures of the study

Participants must also meet at least one of the following conditions:

* Have COVID-19 or COVID-19 like symptoms
* Received a COVID-19 vaccine
* Potential exposure to COVID-19

Exclusion Criteria:

* Unable to provide informed consent
* Unable to perform the requested study tasks and unable or unwilling to assign a proxy informant to complete the tasks

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults living in the US or UK who have COVID-19 or COVID-19 like symptoms, were vaccinated against COVID-19, or were exposed to COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 35278 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
COVID-19 symptom occurrence and severity | 12 months
  Occurrence and severity of potential COVID-19 symptoms as reported by participants in the survey
COVID-19 treatments | 12 months
  Prescription treatments for COVID-19 as reported by participants in the survey
COVID-19 risk factors | 12 months
  Assess potential role of comorbidities and concomitant medications on COVID-19 occurrence and severity
Occurrence and severity of COVID-19 infection after vaccination | 12 months
  Occurrence and severity of COVID-19 infection as reported by participants after SARS-CoV-2 vaccine
Occurrence of medically attended events after vaccination | 1 month
  Occurrence of medically attended events as reported by participants after after SARS-CoV-2 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Dreyer, PhD, MPH, Principal Investigator — Iqvia Pty Ltd
Locations (2):
- IQVIA, Cambridge, Massachusetts, United States
- IQVIA, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that external researchers may want to leverage these data for public health and life sciences research. The intent is to provide limited data access to qualified researchers for research that has gone through a review process.
Supporting Information: Study Protocol
Time Frame: Data will be available during conduct of the study and two years following study completion.
Access Criteria: Qualified researchers that have undergone a review process may submit requests to the IQVIA Registry Data Governance Committee (DGC) requesting approval and access for specific research purposes.

REFERENCES:
- [Derived] Dreyer NA, Knuth KB, Xie Y, Reynolds MW, Mack CD. COVID-19 Vaccination Reactions and Risk of Breakthrough Infections Among People With Diabetes: Cohort Study Derived From Community Reporters. JMIR Diabetes. 2024 Feb 27;9:e45536. doi: 10.2196/45536. PMID 38412008
- [Derived] Largent J, Xie Y, Knuth KB, Toovey S, Reynolds MW, Brinkley E, Mack CD, Dreyer NA. Cognitive and other neuropsychiatric symptoms in COVID-19: analysis of person-generated longitudinal health data from a community-based registry. BMJ Open. 2023 Jun 19;13(6):e069118. doi: 10.1136/bmjopen-2022-069118. PMID 37336535
- [Derived] Reynolds MW, Secora A, Joules A, Albert L, Brinkley E, Kwon T, Mack C, Toovey S, Dreyer NA. Evaluating real-world COVID-19 vaccine effectiveness using a test-negative case-control design. J Comp Eff Res. 2022 Nov;11(16):1161-1172. doi: 10.2217/cer-2022-0069. Epub 2022 Sep 23. PMID 36148919
- [Derived] Reynolds MW, Xie Y, Knuth KB, Mack CD, Brinkley E, Toovey S, Dreyer NA. COVID-19 Vaccination Breakthrough Infections in a Real-World Setting: Using Community Reporters to Evaluate Vaccine Effectiveness. Infect Drug Resist. 2022 Sep 3;15:5167-5182. doi: 10.2147/IDR.S373183. eCollection 2022. PMID 36090603
- [Derived] Dreyer N, Reynolds MW, Albert L, Brinkley E, Kwon T, Mack C, Toovey S. How frequent are acute reactions to COVID-19 vaccination and who is at risk? Vaccine. 2022 Mar 15;40(12):1904-1912. doi: 10.1016/j.vaccine.2021.12.072. Epub 2022 Feb 9. PMID 35177299

DOCUMENTS (1):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04368065/Prot_000.pdf